CLINICAL TRIAL: NCT02758366
Title: An Open-label, Single-arm, Phase II Study to Evaluate Safety and Efficacy of Doxorubicin in Combination With Radiotherapy, Temozolomide and Valproic Acid in Patients With Glioblastoma Multiforme (GBM) and Diffuse Intrinsic Pontine Glioma (DIPG)
Brief Title: Prolonged Exposure to Doxorubicin in Patients With Glioblastoma Multiforme and Diffuse Intrinsic Pontine Glioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to high heterogeneity of enrolled patients
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Iacopo Sardi, MD, PhD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBMTMZ/DOX2015; 2015-002307-28 (EudraCT Number)
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Glioblastoma (GBM); DIPG; Brainstem Glioma, Pediatric; Diffuse Spinal Glioma; Bilateral Thalamic Glioma; Gliomatosis Cerebri; Anaplastic Astrocytoma; Midline Diffuse Glioma
Keywords: glioblastoma multiforme; high grade glioma; diffuse intrinsic pontine glioma; DIPG; doxorubicin; temozolomide; malignant glioma; Brainstem Glioma; diffuse spinal glioma; bilateral thalamic glioma; Anaplastic Astrocytoma; Gliomatosis Cerebri; Midline Diffuse Glioma
MeSH Terms: conditions — Glioblastoma; Neoplasms, Neuroepithelial; Astrocytoma; Glioma; Diffuse Intrinsic Pontine Glioma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin (Experimental): Patients are treated with Weller-Stupp protocol: initial radiotherapy (1.8 Gy/die, days 1-5; total dose 54-60 Gy) with concomitant oral temozolomide (75mg/m2/die, days 1-7) per 6 weeks.
  At week 10 (4 weeks after the chemo-radiotherapy treatment completion): 1 cycle of oral temozolomide (150-180 mg/m2, days 1-5)
  At week 14 (8 weeks after the chemo-radiotherapy treatment completion) 1 cycle of prolonged infusion of Doxorubicin (25mg/m2/die in 24 hours, days 1-4; total cumulative dose 100 mg/m2).
  At week 18 (4 weeks after the end of doxorubicin administration): 16 cycles of oral temozolomide (initial dose of 150 mg/m2 increasing to 180 mg/m2 days 1-5, 28-day cycle).
  Oral valproic acid (20-30 mg/Kg/die bid) is administered from week 1 until the last treatment day.
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin

SUMMARY:
The standard therapy of glioblastoma (GBM) consists of gross total resection followed by focal irradiation to the tumor bed with concomitant and adjuvant temozolomide (TMZ). The association of valproic acid and TMZ during radiotherapy improves survival of GBM. Preclinical studies suggested that doxorubicin had a strong antineoplastic activity against human gliomas. Moreover, some studies showed that the continuous infusion of anthracyclines in patients with solid tumor ensured a better safety profile compared with bolus administration.

Based on these findings, the purpose of this study is to evaluate safety and efficacy of prolonged administration of doxorubicin in combination with radiotherapy, temozolomide and valproic acid in pediatric and adult patients with newly diagnosed GBM and diffuse intrinsic pontine glioma (DIPG).

ELIGIBILITY:
Inclusion Criteria:

* Males and females patients, aged >3 years and < 30 years;
* Newly diagnosed of GBM, DIPG, diffuse brainstem glioma, diffuse spinal glioma, bilateral thalamic glioma, gliomatosis cerebri, anaplastic astrocytoma;
* Patients undergone either surgery or biopsy only;
* No prior chemotherapy and/or radiotherapy;
* Life expectancy ≥ 4 weeks;
* Karnofsky/Lansky ≥ 40 %;
* Written informed consent obtained from the patient/parents or legal representative;
* Adequate hematological function (leucocyte ≥ 2.0 x 10^9/l -Hemoglobin ≥ 10 g/dl - platelet ≥ 50 x 10^9 /l);
* Adequate liver function (total bilirubin ≤ 2.5 x ULN - ALT/AST ≤ 5.0 x ULN);
* Adequate renal function (serum creatinine ≤ 1.5 x ULN);
* Adherence to trial treatment and compliance with the protocol

Exclusion Criteria:

* Any disease or condition that contraindicates the use of the study drug (es. serious mental retardation, brain palsy, congenital syndrome, cardiomyopathy)
* Prior anti-cancer therapy
* Pregnancy or breastfeeding
* Non adequate contraception

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Time to early discontinuation of the study drug (doxorubicin) | 6 months
Number of participants with treatment-related serious adverse events (SAE) as assessed by CTCAE v4.0 | 32 months
  Number of patients with SAE and SAE leading to withdrawal from the study
Number of patients who died for SAE as assessed by CTCAE v4.0 | 32 months
  Mortality due to adverse events
Number of patients who undergone to withdrawal of doxorubicin | 6 months
  Rate of early suspension of the study drug (doxorubicin)

SECONDARY OUTCOMES:
Event free survival | 2 months
  Event free survival (EFS) defined as time (days) between the date of enrolment and the earliest occurence of anyone of the following: progression based on RECIST 1.1 criteria; tumor recurrence; death to any cause.
Overall survival | 2 months
  Overall survival (OS) defined as time between the date of the enrolment and the death to any cause
Progression free survival | 2 months
  Progression free survival (PFS) defined as time between the date of the enrolment and the date tumor progression based on RECIST 1.1criteria
Rate of treatment response | 2 months
  Rate of treatment response (CR, complete response; PR, partial response; SD, stable disease; PD, progressive disease) based on RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital, Florence, Italy

REFERENCES:
- [Background] Eramo A, Ricci-Vitiani L, Zeuner A, Pallini R, Lotti F, Sette G, Pilozzi E, Larocca LM, Peschle C, De Maria R. Chemotherapy resistance of glioblastoma stem cells. Cell Death Differ. 2006 Jul;13(7):1238-41. doi: 10.1038/sj.cdd.4401872. Epub 2006 Feb 3. No abstract available. PMID 16456578
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Ananda S, Nowak AK, Cher L, Dowling A, Brown C, Simes J, Rosenthal MA; Cooperative Trials Group for Neuro-Oncology (COGNO). Phase 2 trial of temozolomide and pegylated liposomal doxorubicin in the treatment of patients with glioblastoma multiforme following concurrent radiotherapy and chemotherapy. J Clin Neurosci. 2011 Nov;18(11):1444-8. doi: 10.1016/j.jocn.2011.02.026. Epub 2011 Aug 2. PMID 21813279
- [Background] Beier CP, Schmid C, Gorlia T, Kleinletzenberger C, Beier D, Grauer O, Steinbrecher A, Hirschmann B, Brawanski A, Dietmaier C, Jauch-Worley T, Kolbl O, Pietsch T, Proescholdt M, Rummele P, Muigg A, Stockhammer G, Hegi M, Bogdahn U, Hau P. RNOP-09: pegylated liposomal doxorubicine and prolonged temozolomide in addition to radiotherapy in newly diagnosed glioblastoma--a phase II study. BMC Cancer. 2009 Sep 2;9:308. doi: 10.1186/1471-2407-9-308. PMID 19725960
- [Background] Cohen KJ, Heideman RL, Zhou T, Holmes EJ, Lavey RS, Bouffet E, Pollack IF. Temozolomide in the treatment of children with newly diagnosed diffuse intrinsic pontine gliomas: a report from the Children's Oncology Group. Neuro Oncol. 2011 Apr;13(4):410-6. doi: 10.1093/neuonc/noq205. Epub 2011 Feb 22. PMID 21345842
- [Background] Krauze AV, Myrehaug SD, Chang MG, Holdford DJ, Smith S, Shih J, Tofilon PJ, Fine HA, Camphausen K. A Phase 2 Study of Concurrent Radiation Therapy, Temozolomide, and the Histone Deacetylase Inhibitor Valproic Acid for Patients With Glioblastoma. Int J Radiat Oncol Biol Phys. 2015 Aug 1;92(5):986-992. doi: 10.1016/j.ijrobp.2015.04.038. Epub 2015 Apr 30. PMID 26194676
- [Background] Lesniak MS, Upadhyay U, Goodwin R, Tyler B, Brem H. Local delivery of doxorubicin for the treatment of malignant brain tumors in rats. Anticancer Res. 2005 Nov-Dec;25(6B):3825-31. PMID 16312042
- [Background] Masoudi A, Elopre M, Amini E, Nagel ME, Ater JL, Gopalakrishnan V, Wolff JE. Influence of valproic acid on outcome of high-grade gliomas in children. Anticancer Res. 2008 Jul-Aug;28(4C):2437-42. PMID 18751431
- [Background] Stan AC, Casares S, Radu D, Walter GF, Brumeanu TD. Doxorubicin-induced cell death in highly invasive human gliomas. Anticancer Res. 1999 Mar-Apr;19(2A):941-50. PMID 10368637
- [Background] van Dalen EC, van der Pal HJ, Caron HN, Kremer LC. Different dosage schedules for reducing cardiotoxicity in cancer patients receiving anthracycline chemotherapy. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD005008. doi: 10.1002/14651858.CD005008.pub3. PMID 19821337
- [Background] Veringa SJ, Biesmans D, van Vuurden DG, Jansen MH, Wedekind LE, Horsman I, Wesseling P, Vandertop WP, Noske DP, Kaspers GJ, Hulleman E. In vitro drug response and efflux transporters associated with drug resistance in pediatric high grade glioma and diffuse intrinsic pontine glioma. PLoS One. 2013 Apr 29;8(4):e61512. doi: 10.1371/journal.pone.0061512. Print 2013. PMID 23637844
- [Background] Weller M, Gorlia T, Cairncross JG, van den Bent MJ, Mason W, Belanger K, Brandes AA, Bogdahn U, Macdonald DR, Forsyth P, Rossetti AO, Lacombe D, Mirimanoff RO, Vecht CJ, Stupp R. Prolonged survival with valproic acid use in the EORTC/NCIC temozolomide trial for glioblastoma. Neurology. 2011 Sep 20;77(12):1156-64. doi: 10.1212/WNL.0b013e31822f02e1. Epub 2011 Aug 31. PMID 21880994